CLINICAL TRIAL: NCT03976011
Title: Validation and Optimization Methods for a Quantitative Characterization of Motion Abnormalities of the Larynx With Echography
Brief Title: Post Thyroidectomy Echographic Method for Study of Vocal Fold Motion
Acronym: VOCALE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: MINDRAY (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K170921J; 2018-A02951-54 (Registry Identifier: IDRCB)
Record Dates: First submitted 2019-05-24; First posted 2019-06-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Laryngeal Nerve Palsy; Postoperative Dysphonia
Keywords: Postoperative dysphonia; Thyroidectomy; Parathyroidectomy; Inferior laryngeal nerve palsy; Trans laryngeal ultrasonography; Quantitative vocal fold motion evaluation; Postoperative recurrent Laryngeal Nerve Palsy
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous Laryngeal Ultrasonography (Experimental): All patients operated on endocrine surgery in the three referral centers and responding to the inclusion criteria will be included after obtaining their writing consent. The gold standard NF will be performed between D1 and D15, as usually performed after these surgeries. TLU will be performed during the same time period by an investigator blind to the NF results. The subject will be his own control, NF and TLU being compared. When facing VF immobility, the subject will benefit from the usual clinical follow up: consultation with NF at 6 weeks and 6 months. TLU will be added to these appointments.
  Interventions: Device: Transcutaneous Laryngeal Ultrasonography

INTERVENTIONS:
Device: Transcutaneous Laryngeal Ultrasonography — TLU will be performed during the same time period of The gold standard NF (who is performed as usually after endocrine surgeries) by an investigator blind to the NF results, between D1 and D15.
  The subject will be his own control, NF and TLU being compared. When facing VF immobility, the subject will benefit from the usual clinical follow up: consultation with NF at 6 weeks and 6 months. TLU will be added to these appointments.

SUMMARY:
One of the major risks of endocrine surgery is recurrent nerve palsy (RNP), leading to vocal folds (VF) immobility. It happens in 5% of cases, leading to high morbidity: dysphonia, aspirations, impossibility to work. Guidelines recommend to systematically perform a nasofibroscopy before and after surgery to check vocal fold mobility. However, due to the decreasing number of specialists, the cost of decontamination, and discomfort of this procedure, these guidelines are insufficiently followed.

Transcutaneous Laryngeal Ultrasonography (TLU) appears a good alternative to nasofibroscopy in evaluating VF mobility, as assessed by the recent flourishing literature. Our team is a leader in this research by having developed a dedicated software, which provides objective measures of VF mobility. The aim of the present protocol is to validate the power of TLU for the diagnosis of RNP on a large cohort of patients operated on endocrine surgery. It is a prospective multicentric study that will blindly compare TLU and nasofibroscopy, the latter being the gold standard. TLU is cost effective and painless; its learning curve is fast. If validated, it may be offered as a good alternative to nasofibroscopy in RNP detection and prognosis.

DETAILED DESCRIPTION:
The rationale of this study is that Transcutaneous Laryngeal Ultrasonography (TLU) may be a relevant and reliable tool in assessing vocal folds (VF) paralysis secondary to endocrine surgery (thyroid and parathyroid surgery). According to the literature and to our own publications, subjective impression of VF (im)mobility seems sufficient to diagnose a paralysis. However, the investigators think that objective measures, based on a dedicated semi-automatic software, may offer a much powerful implement and needs to be compared to the gold standard technique, i.e. the nasofibroscopy (NF), in a large prospective multicentric cohort.

In a preliminary study, the investigators described TLU anatomical landmarks first in an ex vivo study and secondary in a prospective study based on 50 patients with VF paralysis compared to 50 controls. These three landmarks, the two arytenoids and the anterior insertion of the two vocal folds on the thyroid cartilage, are easy to recognize, and independent of the postoperative delay and the person performing TLU. They define two symmetrical hemi-larynges in healthy subjects. The investigators designed an original software, aiming at offering two quantitative criteria of laryngeal mobility and symmetry, taking into account motion symmetry (symmetry index) and amplitude (mobility index) of the two hemi-larynges. When a subject presented with a unilateral VF paralysis, the mean symmetry index was significantly larger compared to the control group (20.4% ±13.8% versus 6.7% ±4.7%, p<0.0001) and the mean lower mobility index was significantly smaller (2.2% ±17.4% versus 20.5% ±14.8%, p<0.0001). The sensitivity and specificity of this first version of our automatized protocol were 82%.

The aim of the present study is to validate TLU as an alternative to NF in a large independent cohort of patients operated on endocrine surgery. The main goal is to improve the sensitivity and specificity of the objective measures and implement new parameters in the software. By a ready to use tool, the investigators would like to offer the opportunity to any practitioner to assess and quantify VF (im)mobility with their usual US machine.

The subjects will be recruited in the three different clinical centers, highly specialized in endocrine surgery. The aim of 500 subjects included seems feasible thanks to the high activity of these centers. Moreover the latter already have sufficient and qualified staff and technical tools to perform clinical follow up, US, and NF.

The technical acquisition is as follow. The TLU is performed with a 7-14 MHz linear probe, using a portable machine. Subjects are lying on the back, neck slightly extended, with the probe placed over the laryngeal prominence of the thyroid cartilage, including the arytenoids in the axial view. The images are acquired in B-mode, during normal breathing at rest. Typical values for acquisition are: frequency 10 MHz, depth of field of view 4 cm, mechanical index 0.6, gain 45%, dynamic range 85 decibels. A video clip of 10 seconds (30 images per second) is recorded in order to include 5 to 6 complete respiratory cycles. Two images corresponding to physiological abduction and adduction during the same breath cycle are selected. The landmarks, previously described, are selected on the images and tracked by the software.

All patients operated on endocrine surgery in the three referral centers and responding to the inclusion criteria will be included after obtaining their writing consent. The gold standard NF will be performed between D1 and D15, as usually performed after these surgeries. TLU will be performed during the same time period by an investigator blind to the NF results. The subject will be his own control, NF and TLU being compared. When facing VF immobility, the subject will benefit from the usual clinical follow up: consultation with NF at 6 weeks and 6 months. TLU will be added to these appointments.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old patient and older
2. Free informed consent of the patient obtained during the preoperative consultation or, failing this, the day before the intervention during the preoperative hospitalization
3. Thyroid / parathyroid surgery scheduled within 3 months, regardless of the indication or extension
4. Affiliation to a social security system (recipient or assign) excluding AME.

Exclusion criteria

1. Known preoperative history of recurrent nerve palsy
2. History of thyroid or parathyroid surgery or cervicotomy for another pathology
3. History of laryngeal tumor or vocal folds
4. Patient under guardianship or curatorship or deprived of liberty or under judicial protection
5. Pregnant, breastfeeding and parturient women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance associated with the postoperative quantitative TLU (i.e. measured by asymmetry in vocal cord mobility obtained with our dedicated software of image analysis) for the diagnostic of postoperative recurrent nerve palsy (RNP). | Between Day 1(the day after the surgery) and Day 15
  The diagnostic performance of the postoperative measurement of asymmetry in vocal cord mobility obtained with the quantitative TLU will be evaluated by the area under the roc curve and its 95% confidence interval. The gold standard for diagnosis of postoperative RNP will be the nasofibroscopy performed between Day 1 and Day15.

SECONDARY OUTCOMES:
Diagnostic performance associated with the postoperative qualitative TLU (i.e. obtained by the operator during TLU, without the use of our dedicated software for the diagnostic of postoperative recurrent nerve palsy (RNP). | Between Day 1(the day after the surgery) and Day 15
  The diagnostic performance of the postoperative qualitative evaluation of asymmetry in vocal cord mobility obtained by the operator during TLU will be evaluated using sensitivity, specificity, positive and negative predictive value and and their 95% confidence interval. The gold standard for diagnosis of postoperative RNP will be the nasofibroscopy performed between Day 1 and Day 15.
Predictive performance associated with the postoperative quantitative TLU for the diagnosis of final recovery of RNP, among subjects with postoperative RNP. | 6 months after surgery
  The predictive performance of the measurement of asymmetry in vocal cord mobility obtained with the postoperative quantitative TLU will be evaluated among patients with postoperative RNP by the area under the roc curve and its 95% confidence interval. The gold standard for diagnosis of final recovery of RNP will be the nasofibroscopy performed 6 months after surgery.
Predictive performance associated with the postoperative qualitative TLU for the diagnosis of final recovery of RNP, among subjects with postoperative RNP. | 6 months (e.g. 6 months after surgery)
  The predictive performance of the postoperative qualitative evaluation of asymmetry in vocal cord mobility obtained by the operator during TLU will be evaluated using sensitivity, specificity, positive and negative predictive value and and their 95% confidence interval. The gold standard for diagnosis of final recovery of RNP will be the nasofibroscopy performed 6 months after surgery.
Predictive performance associated with the quantitative TLU performed 6 weeks after surgery for the diagnosis of final recovery of RNP, among subjects with postoperative RNP. | 6 months after surgery
  The predictive performance of the measurement of asymmetry in vocal cord mobility obtained with the quantitative TLU 6 weeks after surgery will be evaluated among patients with postoperative RNP by the area under the roc curve and its 95% confidence interval. The gold standard for diagnosis of final recovery of RNP will be the nasofibroscopy performed 6 months after surgery.
Predictive performance associated with the qualitative TLU performed 6 weeks after surgery for the diagnosis of final recovery of RNP, among subjects with postoperative. | 6 months after surgery
  The predictive performance of the qualitative evaluation of asymmetry in vocal cord mobility obtained by the operator during TLU performed 6 weeks after surgery will be evaluated using sensitivity, specificity, positive and negative predictive value and and their 95% confidence interval. The gold standard for diagnosis of final recovery of RNP will be the nasofibroscopy performed 6 months after surgery.
Diagnostic performance associated with the quantitative TLU performed 6 months after surgery for the diagnosis of final recovery of RNP, among subjects with postoperative RNP. | 6 months after surgery
  The diagnostic performance of the measurement of asymmetry in vocal cord mobility obtained with the quantitative TLU 6 months after surgery will be evaluated among patients with postoperative RNP by the area under the roc curve and its 95% confidence interval. The gold standard for diagnosis of final recovery of RNP will be the nasofibroscopy performed 6 months after surgery.
Diagnostic performance associated with the qualitative TLU performed 6 months after surgery for the diagnosis of final recovery of RNP, among subjects with postoperative RNP. | 6 months after surgery
  The diagnostic performance of the qualitative evaluation of asymmetry in vocal cord mobility obtained by the operator during TLU performed 6 months after surgery will be evaluated using sensitivity, specificity, positive and negative predictive value and and their 95% confidence interval. The gold standard for diagnosis of final recovery of RNP will be the nasofibroscopy performed 6 months after surgery.
Correlation between the postoperative Voice Handicap Index (VHI) and the postoperative quantitative TLU. | Between Day 1(the day after the surgery) and Day 15
  Pearson correlation coefficient between postoperative quantitative TLU and VHI
Correlation between the Voice Handicap Index (VHI) measured 6 weeks after surgery and the quantitative TLU measured 6 weeks after surgery, among subjects with postoperative RNP. | 6 weeks after surgery (+/- 15 days)
  Pearson correlation coefficient between quantitative TLU and VHI at 6 weeks
Correlation between the Voice Handicap Index (VHI) measured 6 months after surgery and the quantitative TLU measured 6 months after surgery, among subjects with postoperative RNP. | 6 months after surgery
  Pearson correlation coefficient between quantitative TLU and VHI at 6 months
Pearson correlation coefficient between postoperative quantitative TLU and loss or diminution of the intraoperative stimulation of the inferiors laryngeal nerves, expressed in microvolts, measured during the surgery. | Between Day 1(the day after the surgery) and Day 15
Postoperative patient's satisfaction regarding TLU examination: six-point satisfaction questionnaire | Between Day 1 and Day 15
  Patient's satisfaction regarding TLU examination will be evaluated using a structured questionnaire (Strongly disagree; Slightly disagree; Neither agree nor disagree; Slightly agree; Strongly agree; Without opinion)
Postoperative patient's satisfaction regarding nasofibroscopic examination: six-point satisfaction questionnaire | Between Day 1 and Day 15
  Postoperative patient's satisfaction regarding nasofibroscopic examination will be evaluated using a structured six-point satisfaction six-point satisfaction questionnaire (Strongly disagree; Slightly disagree; Neither agree nor disagree; Slightly agree; Strongly agree; Without opinion)
Comparison between the costs associated with the nasofibroscopy of the one hand, and the TLU on the other hand. | 6 months
  The costs of nasofibroscopy on the one hand, and the TLU on the other, will be determined taking into account of the french social security system and its repayment as well as the time required to carry out the examinations, the purchase cost of the devices and its maintenance. The costs associated with the two examinations will be compared using the incremental cost-effectiveness ratio (ICER) and its 95% confidence interval

OTHER OUTCOMES:
Diagnostic performance associated with the postoperative measurements obtained with the interactive software developed by the Mindray company of different points of the laryngeal anatomy for the diagnostic of postoperative recurrent nerve palsy (RNP). | Between Day 1 (the day after the surgery) and D15
  The diagnostic performance of the postoperative measurement of asymmetry in vocal cord mobility obtained with the interactive software developed by the Mindray company will be evaluated by the area under the roc curve and its 95% confidence interval. The gold standard for diagnosis of postoperative RNP will be the nasofibroscopy performed between Day 1 and Day 15.
Diagnostic performance comparison of the postoperative measure obtained with an interactive software developed by the Mindray company and with quantitative TLU measured by asymmetry in vocal cord mobility with our dedicated software of image analysis. | Between Day 1 (the day after the surgery) and Day 15
  Comparison between the area under the roc curve of these two measurements, using Delong test.
Concordance between the postoperative measure obtained with an interactive software developed by the Mindray company and with quantitative TLU (i.e. measured by asymmetry in vocal cord mobility obtained with our dedicated software of image analysis). | Between Day 1 (the day after the surgery) and Day 15
  The concordance between these two measurements will be evaluated using a Bland and Altman plot

CONTACTS AND LOCATIONS:
Overall Officials: Christophe TRESALLET, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - CHU Nantes - Clinique de chirurgie Digestive et Endocrinienne, Nantes
  - Hopital Pitié-Salpêtrière, Paris
  - Hopital Avicenne, Paris
  - Hopital Cochin, Paris
  - Institut Gustave Roussy (IGR), Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergeret-Cassagne H, Lazard DS, Lefort M, Hachi S, Leenhardt L, Menegaux F, Russ G, Tresallet C, Frouin F. Sonographic Dynamic Description of the Laryngeal Tract: Definition of Quantitative Measures to Characterize Vocal Fold Motion and Estimation of Their Normal Values. J Ultrasound Med. 2017 May;36(5):1037-1044. doi: 10.7863/ultra.16.05014. Epub 2017 Jan 10. PMID 28072470
- [Background] Lazard DS, Bergeret-Cassagne H, Lefort M, Leenhardt L, Russ G, Frouin F, Tresallet C. Transcutaneous Laryngeal Ultrasonography for Laryngeal Immobility Diagnosis in Patients with Voice Disorders After Thyroid/Parathyroid Surgery. World J Surg. 2018 Jul;42(7):2102-2108. doi: 10.1007/s00268-017-4428-2. PMID 29299645